CLINICAL TRIAL: NCT02117947
Title: Behavioral Counseling to Reduce Children's Secondhand Smoke Exposure: A Trial With Maternal Smokers
Brief Title: Counseling to Reduce Children's SHS Exposure: A Trial With Maternal Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01CA105183 (NIH); R01CA105183 (NIH)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Nicotine Dependence
Keywords: child secondhand smoke; maternal smoking; tobacco; nicotine; behavioral counseling; low-income; underserved
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Counseling (Experimental): Behavioral counseling used evidence-based smoking cessation intervention components as well as a theoretically-framed focus on behavioral shaping to promote the adoption of smoke-free homes and cars. Sessions included two, 1-hour in-home counseling and seven, 5-15 minute telephone follow-up sessions over 16 weeks. Content included health ed around the benefits of eliminating children's exposure to secondhand smoke; skills training around adoption and maintenance of smoke-free environments; goal setting, problem solving, and positive reinforcement for progress toward goals; coping skills training for smoking urge and mood management; and home support for maternal smoking behavior change achieve through family contracts and home detailing promoting pro-smoke-free home norms.
  Interventions: Behavioral: Behavioral Counseling
- Self-help control (Active Comparator): The self-help control group received a comprehensive self-help manual that outlined all of the goals and strategies covered in counseling, however, counseling was not provided to this group.
  Interventions: Behavioral: Self-help control

INTERVENTIONS:
Behavioral: Behavioral Counseling — Behavioral counseling used components of evidence-based smoking intervention treatment to promote maternal smokers efforts in reducing their children's exposure to secondhand smoke.
  Arms: Behavioral Counseling
Behavioral: Self-help control — This intervention group received a comprehensive self-help manual that included information and advice about how to protect children from secondhand smoke (e.g., adopting a smokefree home and car.)
  Arms: Self-help control

SUMMARY:
The goal of this study is to reduce infant and toddlers' secondhand smoke exposure (SHSe) in a high risk, medically underserved population of maternal smokers. The program is called "Philadelphia FRESH (Family Rules for Establishing Smokefree Homes)". Participants are recruited from low-income urban neighborhoods in Philadelphia, Pennsylvania. After determining study eligibility via telephone screen, all participants complete an in-home pre-intervention interview that includes self-reported smoking history, current smoking and exposure patterns, and factors that relate to maternal smoking (such as depressive symptoms, weight concerns, nicotine dependence,) as well as collection of child urine cotinine (a biomarker used to detect SHSe).

Participants are randomized after baseline to receive either (a) a moderately intensive (up to 2 in-home sessions, 8 phone sessions) Behavioral Counseling intervention (BC) delivered over a 16-week period by counselors trained and supervised by investigators, or (b) an enhanced Self-Help Control (SHC) that uses brief advice and a detailed self-help manual for SHSe-reduction and smokingcessation. Post intervention assessments include self-reports of intervention process, factors associated with intervention effects, and intervention outcomes that include child urine cotinine (to measure level of SHSe) and participant saliva cotinine (to verify self-reported smoking quit status). Interviewers and data management staff remain blind to the treatment assignment. All procedures are implemented after signed informed consent and were approved by Temple University's Institutional Review Board.

DETAILED DESCRIPTION:
This study represents a community-based behavioral counseling trial designed to reduce infant and toddlers' secondhand smoke exposure (SHSe) in a high risk, medically underserved population of African American maternal smokers. The program is called "Philadelphia FRESH (Family Rules for Establishing Smokefree Homes)". Participants are recruited from low-income urban neighborhoods in Philadelphia, Pennsylvania via posters on mass transit, newspaper ads, and referral from pediatricians or community WIC clinics.

Inclusion Criteria:

* mothers who smoke at least 5 cigarettes per day
* have a child under 4 years of age
* report exposing their youngest child to at least 2 of her cigarettes per day. (Child exposure to a cigarette is defined as a child being in the same room or car when adult is smoking. Room is defined as 4-walls and a door that closes.)

Exclusion Criteria:

* Diagnosis of a Axis I psychiatric disorder
* pregnant
* not proficient in English.

After determining study eligibility via telephone screen, all participants complete an in-home baseline interview that includes self-reported smoking history, current smoking and exposure patterns, and factors that relate to maternal smoking (such as depressive symptoms, weight concerns, nicotine dependence,) as well as collection of child urine cotinine (a biomarker used to detect SHSe).

Participants are randomized to receive either a Behavioral Counseling intervention (BC) delivered over a 16-week period by master's level counselors trained and supervised by PhD-level investigators, or an enhanced Self-Help Control (SHC) that uses a detailed self-help manual for SHSe-reduction and smoking cessation. Post intervention assessments at 16 weeks, 3- and 12-month follow-up include self-reports of factors associated with intervention effects and intervention outcomes that include child urine cotinine (to measure level of SHSe) and participant saliva cotinine (to verify self-reported smoking quit status). Interviewers and data management staff remain blind to the treatment assignment. All procedures are implemented after signed informed consent and were approved by Temple University's Institutional Review Board.

Behavioral Counseling (BC): Mothers randomized to receive BC complete two in-home, and up to a 8 proactive telephone counseling sessions within a 16-week period. Mothers also receive four health education and self-help mailings sent in two week intervals during the first 8 weeks of their participation to supplement the counseling content. (These four mailings are identical to the self-help materials received by the control group.) The overarching goal of child SHSe reduction is intended to be achieved through specific BC objectives. These objectives include facilitation of health education regarding the dangers of SHSe and smoking, plus the benefits of SHSe-reduction and smoking cessation to maternal and child health. Additional objectives include (a) building family-level social support to facilitate home-level smoking behavior change; (b) fostering coping and problem-solving skills to help participants manage smoking urges as well as general life stressors; (c) providing and modeling abundant positive reinforcement following SHSe reduction efforts to facilitate confidence and motivation for more challenging smoking behavior change goals.

Self-Help Control (SHC) group: Participants in SHC group receive an intervention binder with brief advice by telephone on how to use the manual for SHSe reduction. The binder contains information identical to the BC group, however, all binder content is included in this single mailing.

Primary study outcomes include change in (a) maternal-reported child SHSe (reported as cigarettes exposed per day) obtained via validated timeline follow-back methods; and (b) baby urine cotinine- a biomarker of SHSe standard in tobacco exposure studies. Secondary outcomes include (a) change in maternal cigarettes smoked per day and (b) maternal reported 7-day point prevalence abstinence, bioverified by saliva cotinine. Urine and saliva samples were assayed for cotinine using high performance liquid chromatography-tandem mass spectrometry as an indicator of exposure to tobacco smoke.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who smoke at least 5 cigarettes per day
* have at least one child under 4 years of old (youngest child is target child for data collection (urine cotinine)
* report exposing youngest (target) child to at least 2 of her cigarettes/day (defined as child in the same room [4-walls and a door that closes] or car when someone is actively smoking a cigarette.

Exclusion Criteria:

* current diagnosis or treatment of a psychiatric disorder
* currently pregnant
* not proficient in English

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
child urine cotinine | baseline to 16 weeks
  tobacco exposure biomarker measured in n/mL

SECONDARY OUTCOMES:
maternal reported child tobacco smoke exposure | baseline to 16 weeks
  7-day point prevalence cigarettes per day exposed
maternal reported smoking | baseline - 16 weeks
  7 day point prevalence cigarettes smoked per day
maternal smoking abstinence | baseline to 16 weeks
  7-day cotinine-verified point prevalence abstinence

OTHER OUTCOMES:
post-treatment maternal reported child tobacco smoke exposure | 3- and 12-month post treatment follow-up
  7-day point prevalence cigarettes per day exposed
post-treatment child cotinine | 3- and 12-month post treatment follow-up
  tobacco exposure biomarker measured in n/mL
post-treatment maternal smoking abstinence | 3- and 12-month post treatment follow-up
  7-day cotinine-verified point prevalence abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Bradley N Collins, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University Health Behavior Research Clinic, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collins BN, Wileyto EP, Hovell MF, Nair US, Jaffe K, Tolley NM, Audrain-McGovern J. Proactive recruitment predicts participant retention to end of treatment in a secondhand smoke reduction trial with low-income maternal smokers. Transl Behav Med. 2011 Sep;1(3):394-9. doi: 10.1007/s13142-011-0059-6. PMID 24073063
- [Background] Collins BN, Nair U, Hovell MF, Audrain-McGovern J. Smoking-related weight concerns among underserved, black maternal smokers. Am J Health Behav. 2009 Nov-Dec;33(6):699-709. doi: 10.5993/ajhb.33.6.7. PMID 19320618
- [Background] Collins BN, Ibrahim JK, Hovell M, Tolley NM, Nair US, Jaffe K, Zanis D, Audrain-McGovern J. Residential smoking restrictions are not associated with reduced child SHS exposure in a baseline sample of low-income, urban African Americans. Health (Irvine Calif). 2010 Nov;2(11):1264-1271. doi: 10.4236/health.2010.211188. PMID 23875066
- [Background] Collins BN, Ibrahim J. Pediatric Secondhand Smoke Exposure: Moving Toward Systematic Multi-Level Strategies to Improve Health. Glob Heart. 2012 Jul;7(2):161-165. doi: 10.1016/j.gheart.2012.05.001. No abstract available. PMID 24040587
- [Background] Collins BN, Nair US, Shwarz M, Jaffe K, Winickoff J. SHS-Related Pediatric Sick Visits are Linked to Maternal Depressive Symptoms among Low-Income African American Smokers: An Opportunity for Intervention in Pediatrics. J Child Fam Stud. 2013 Oct;22(7):1013-21. doi: 10.1007/s10826-012-9663-4. PMID 24339721
- [Background] Shwarz M, Collins BN, Nair US. Factors associated with maternal depressive symptoms among low-income, African American smokers enrolled in a secondhand smoke reduction programme. Ment Health Fam Med. 2012 Dec;9(4):275-87. PMID 24294302
- [Background] Collins BN, DiSantis KI, Nair US. Longer previous smoking abstinence relates to successful breastfeeding initiation among underserved smokers. Breastfeed Med. 2011 Dec;6(6):385-91. doi: 10.1089/bfm.2010.0076. Epub 2011 Jan 21. PMID 21254795
- [Background] Collins BN, Levin KP, Bryant-Stephens T. Pediatricians' practices and attitudes about environmental tobacco smoke and parental smoking. J Pediatr. 2007 May;150(5):547-52. doi: 10.1016/j.jpeds.2007.01.006. PMID 17452234
- [Derived] Collins BN, Nair US, DiSantis KI, Hovell MF, Davis SM, Rodriguez D, Audrain-McGovern J. Long-term Results From the FRESH RCT: Sustained Reduction of Children's Tobacco Smoke Exposure. Am J Prev Med. 2020 Jan;58(1):21-30. doi: 10.1016/j.amepre.2019.08.021. Epub 2019 Nov 21. PMID 31759804
- [Derived] Collins BN, Nair US, Davis SM, Rodriguez D. Increasing Home Smoking Restrictions Boosts Underserved Moms' Bioverified Quit Success. Am J Health Behav. 2019 Jan 1;43(1):50-56. doi: 10.5993/AJHB.43.1.5. PMID 30522566
- [Derived] Collins BN, Nair US, Hovell MF, DiSantis KI, Jaffe K, Tolley NM, Wileyto EP, Audrain-McGovern J. Reducing Underserved Children's Exposure to Tobacco Smoke: A Randomized Counseling Trial With Maternal Smokers. Am J Prev Med. 2015 Oct;49(4):534-44. doi: 10.1016/j.amepre.2015.03.008. Epub 2015 May 28. PMID 26028355